CLINICAL TRIAL: NCT01535599
Title: Safety and Efficacy Evaluation of Topical AL-60371 Otic Suspension, 0.3% in the Treatment of Acute Otitis Externa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-10-018
Record Dates: First submitted 2012-02-15; First posted 2012-02-20 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-06

CONDITIONS: Acute Otitis Externa
Keywords: Acute Otitis Externa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AL-60371 (Experimental): AL-60371, 0.3% Otic Suspension, 4 drops to the affected ear(s) twice daily for 7 days
  Interventions: Drug: AL-60371, 0.3% Otic Suspension
- Vehicle (Placebo Comparator): AL-60371 Vehicle, 4 drops to the affected ear(s) twice daily for 7 days
  Interventions: Other: AL-60371 Vehicle

INTERVENTIONS:
Drug: AL-60371, 0.3% Otic Suspension
  Arms: AL-60371
Other: AL-60371 Vehicle — Inactive ingredients used as a placebo comparator
  Arms: Vehicle

SUMMARY:
The purpose of this study was to demonstrate the superiority of AL-60371, 0.3% Otic Suspension relative to AL-60371 Vehicle based on clinical cures at test-of-cure (TOC) for the treatment of acute otitis externa (AOE).

DETAILED DESCRIPTION:
Patients were evaluated for safety and efficacy during the visits conducted at Day 3 (on-therapy), Day 8 (end-of-therapy), and Day 11 (TOC). Patients or parents/legal guardians completed a telephone diary twice daily to record assessments of ear pain, ear pain medication use, and the impact of ear pain on sleep and other daily activities.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months of age.
* Clinical diagnosis of acute otitis externa (AOE) based on clinical observation and of presumed bacterial origin in at least one ear.
* Combined numerical score of ≥4 in at least one affected ear at the Day 1 exam for tenderness, erythema, and edema.
* Agree to refrain from water immersion of the ears during the conduct of the entire study.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Duration of signs or symptoms of AOE greater than 28 days in the affected ear(s) as reported by patient or parent/guardian.
* Presence of a tympanostomy tube or perforated tympanic membrane in the affected ear(s).
* Clinically diagnosed otic disease other than AOE (eg, malignant otitis externa) in the affected ear(s).
* Known or suspected ear infection of yeast, fungal or mycobacterial origin in the affected ear(s).
* Prior otologic surgery within 6 months of study entry in the affected ear(s).
* Known or suspected allergy or hypersensitivity to quinolones or other ingredients present in the medications to be used in the study.
* Patients who use ear plugs, head phones or ear buds and are unwilling to discontinue their use during the study period.
* Other protocol-defined exclusion criteria may apply.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 768 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sally Scheib, Sr. Clinical Project Lead, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 68 investigational centers located in the United States, Puerto Rico, and Canada.
Pre-assignment Details: Of the 768 consented participants, 75 were exited from the study as screen failures prior to randomization. This reporting group includes all randomized participants (693).
Period: Overall Study
Arm/Group | AL-60371 | Vehicle
Started | 347 | 346
Completed | 297 | 250
Not Completed | 50 | 96
Not completed — Adverse Event | 6 | 15
Not completed — Lost to Follow-up | 3 | 4
Not completed — Subj Decision Unrelated to Adverse Event | 4 | 3
Not completed — Treatment Failure | 33 | 66
Not completed — BL Culture + for Group A Strep | 0 | 1
Not completed — BL Culture + for Yeast//Fungi | 0 | 1
Not completed — Randomized in Error | 2 | 4
Not completed — Did not use product | 1 | 0
Not completed — Other | 1 | 0
Not completed — Stopped medication | 0 | 1
Not completed — Noncompliance | 0 | 1

BASELINE CHARACTERISTICS:
Population: This reporting group includes all randomized participants who were treated with study medication (686). Note: 6 participants were randomized in error and did not receive study medication (3 in AL-60371 and 3 in Vehicle). Additionally 1 participant randomized to Vehicle exited the study at Visit 2 without dosing the study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | AL-60371 | Vehicle | Total
Number analyzed (Participants) | 344 | 342 | 686
Age, Customized [Number; unit: participants]
  Infants/Toddlers (18 days to 23 months) | 3 | 2 | 5
  Children (2 to 11 years) | 61 | 83 | 144
  Adolescents (12 to 17 years) | 64 | 42 | 106
  Adults (18 to 64 years) | 195 | 186 | 381
  Elderly (≥ 65 years) | 21 | 29 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 183 | 385
  Male | 142 | 159 | 301

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Clinical Cures at the Day 11 (TOC) Visit
Description: An otoscopic exam was conducted by the physician. Clinical cure was considered attained if the sum of the numerical scores of the 3 signs and symptoms of AOE (tenderness, erythema, and edema) was 0 at Day 11. In this analysis, the clinical cure outcome at Day 11 (TOC) was considered a failure for all pathogen positive patients who did not complete the study (for any reason). Proportion of patients is reported as a percentage.
Time Frame: Day 11
Population: This analysis population includes the pathogen positive participants of the intent-to-treat (ITT) analysis set, ie, all participants who received study medication and were pathogen positive in the study ear at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | AL-60371 | Vehicle
Number analyzed (Participants) | 145 | 138
percentage of participants | 71.7 | 33.3

2. Secondary Outcome: Proportion of Patients With Microbiological Successes at the Day 11 (TOC) Visit
Description: Microbiological success was considered attained if all pretherapy bacteria were absent from the exit otic specimen. The presence of fungi and/or yeast was not considered in the determination of microbiological success. In this analysis, the microbiological success value at Day 11 (TOC) was considered a failure for all pathogen positive patients who did not complete the study (for any reason). Proportion of patients is reported as a percentage.
Time Frame: Day 11
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | AL-60371 | Vehicle
Number analyzed (Participants) | 145 | 138
percentage of participants | 66.9 | 13.0

3. Secondary Outcome: Median Time to Cessation of Ear Pain as Reported by the Patient or Parent/Legal Guardian Via the Telephone Diary
Description: Cessation of ear pain was defined as occurring on the first time point that ear pain was absent (morning or evening) and did not return in any subsequent diary entries. Day 1 was the starting point for this time-to-event analysis. For this analysis, all patients who did not complete the study and ear pain never ceased had their ear pain considered as being present throughout the planned duration of the study.
Time Frame: Time to event, up to Day 11
Population: This analysis population includes the pathogen positive participants of the intent-to-treat (ITT) analysis set, ie, all participants who received study medication and were pathogen positive in the study ear at baseline. Patients who did not report ear pain at any diary entry during first 7 days of the study were excluded from the analysis.
Measure: Median (Standard Error); unit: days
Arm/Group | AL-60371 | Vehicle
Number analyzed (Participants) | 138 | 128
days | 4.0 (0.2) | 7.0 (0.4)

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected for the duration of the study (1 year, 2 months). An AE was considered to be any untoward medical occurrence in a participant who was exposed to the study medication, regardless of causal relationship.
Description: This reporting group includes all randomized participants who were treated with study medication (686). AEs were obtained as solicited comments from the study participants and as observations by the study Investigator.
Arm/Group | AL-60371 | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/344 | 1/342
Other Adverse Events (participants affected / at risk) | 0/344 | 0/342
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AL-60371 (N=344) | Vehicle (N=342)
Anxiety (Psychiatric disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.